CLINICAL TRIAL: NCT06804395
Title: CanScan; Community-based Registry to Assess, Address and advaNce SCreening for cANcer Prevention and Management
Status: Recruiting | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: Pro2024-0211
Record Dates: First submitted 2025-01-17; First posted 2025-02-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cancer Risk
Keywords: Cancer Prevention; Cancer Risk; Cancer Early Detection; Cancer High Risk

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early diagnosis of cancer allows for better treatment outcomes, higher survival rates, and lower costs of care. It is shown that cancer monitoring for cancer in at-risk populations is a key component in early diagnosis. The HMH Hennessey Institute for Cancer prevention and Applied Molecular Science (HICAP) is a newly founded institute, providing clinical services for cancer screening and risk assessment to the community, as well as research in cancer risk and prevention. The CanScan registry will prospectively collect data from participants in the form of questionnaires. The registry will also capture data that is collected as per non-research assessments, for participants who consent to participate. The registry will facilitate better understanding of cancer risk, screening, and diagnostics.

ELIGIBILITY:
* Adults ( 18 and older)
* Ability to provide own consent
* Must meet at least one of the below criteria, Indicating an increased risk for cancer, any of the following:

  * Family or personal history suggests a familial/hereditary disorder known or suspected of predisposition to cancer.
  * Personal factors associated with an increased risk for cancer include benign breast disease, polyps, tobacco use, etc.as defined by the investigator.
  * Family members of participating individuals.
* Any participant in the HICAP program regardless of cancer risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are at risk for cancer or who have taken the Hennessy Institute cancer risk assessment (I.e participated in their cancer prevention program)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2034-10-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Pathogenic Germline Variants (PGV) | 10 years from study initiation as defined based on the date the first patient was enrolled.
  Compare the number of detected PGVs as measured by a universal multi-gene panel, proactively, in a diverse community-based population of individuals. PGV rate will be compared to NCCN genetic testing criteria at baseline, and to longitudinal cancer outcomes.

SECONDARY OUTCOMES:
Incidence of Cancer | 10 years from study enrollment.
  The number of new cancer cases diagnosed in participants with specific PGV's (i.e. "at high risk" to develop cancer) compared to those without these markers (i.e. "low / average risk") over a period of ten years as described below.
Genetic Risk Score (GRS) | 10 years from study enrollment
  GRS is a score that includes demographic data, Family history, Medical history, Epidemiologic risk factors and data stemming from SOC biospecimens analysis. The purpose of this is to assess the association between PGV's, GRS's and the time to cancer diagnosis.
Environmental and Lifestyle Factors | 10 years from study enrollment
  We will evaluate the interaction between genetic markers and environmental/lifestyle factors (e.g., smoking, diet, physical activity) on cancer risk. This will be achieved by assessing environmental/lifestyle factors via questionnaires and correlating these with cancer incidence (Secondary Outcome 2)
Impact of Early Detection and Prevention on Cancer Outcomes | 10 years from study enrollment
  This study will evaluate the association between various preventive measures (e.g., regular screenings, lifestyle modifications) as reported via questionnaires and cancer outcomes (defined as overall survival, and disease-free survival).

CONTACTS AND LOCATIONS:
Overall Officials: Elias Obeid, MD, MPH, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hennessy Institute for Cancer Prevention and Applied Molecular Medicine, Totowa, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided